CLINICAL TRIAL: NCT02536599
Title: Risk Factors & Outcomes for Clinically Documented Infections in Pediatric Cancer Patients With Fever & Neutropenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Doc Inf FN Ped Onc
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Febrile Neutropenia
Keywords: Febrile Neutropenia; Childhood Cancer; Pediatric Oncology; Fever; Neutropenia
MeSH Terms: conditions — Febrile Neutropenia; Neoplasms; Fever; Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to identify clinical and laboratory parameters, present at the time of initial evaluation that could help predict which children with cancer, fever, and neutropenia will be at risk for developing clinically documented infections and/ or complications.

DETAILED DESCRIPTION:
Background:

It has long been recognized that not all neutropenic patients have the same risk of developing serious infections and/or complications.

Fever and infection represent the most important complications of myeloablative cytotoxic therapy that results in severe mucositis and prolonged neutropenia .

One of the most important concepts in the approach to infections in the febrile neutropenic patient is the recognition of risk. Risk can be defined in two ways. First, risk may be defined in terms of the probability for developing a febrile neutropenic infection; and second, it may be defined in terms of the likelihood for significantly poor outcomes due to that infection.

An understanding of the risks in the latter case may be used to define the approaches to management; for instance, in-patient versus out-patient treatment strategies and administration of intravenous versus oral formulations of antimicrobial therapy. These considerations have significant economic and quality of life ramifications.

Many institutions have developed simple clinical criteria to identify low-risk patients without having to calculate a risk-index score. This might be a more practical method in busy clinical settings, or as a tool in setting of low resource country.

Patients & Methods:

The study will include children, either referred from the pediatric oncology clinic, or who have been previously admitted to the pediatric oncology department, those who have been documented with episodes of fever and neutropenia at South Egypt Cancer Institute (SECI), and fulfilling all criteria for enrollment in this study.

All the patients at the time of initial evaluation will be subjected to complete clinical history and full clinical examination.

The enrolled patients will be followed for either developing clinically evident infection e.g., pneumonia, gastroenteritis, meningitis, septicemia, etc.), or until resolution of fever and/ or neutropenia. The risk for either developing clinically evident infection, or not, will be assessed according to clinical and laboratory parameters, present at the time of initial evaluation to identify those patients who would be more prone to develop infection and/ or complications Fever is defined as a temperature greater than or equal to 38.3 C occurring once or a temperature greater than or equal to 38 C occurring twice during a 24-hour period.

Patients with an absolute neutrophilic count (ANC) of less than 500/mm3 and those with an ANC of less than 1,000/mm3 and decreasing will be considered neutropenic.

Complete blood count & other diagnostic studies, including laboratory studies and imaging procedures will be obtained if needed to further evaluate and determine the source of fever and/or infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years.
* Patients diagnosed with hematologic malignancies or solid tumors.
* Patients admitted at the pediatric oncology department for at least 24-hour period after documentation of an episode of fever & neutropenia at the time of initial evaluation at the pediatric oncology clinic.
* Patients who previously have been admitted at the pediatric oncology department, after documentation of an episode of fever & neutropenia.

Exclusion Criteria:

* Patients whose age is more than 18 years.
* Patients not fulfilling the criteria for diagnosis of fever and neutropenia.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients who have episodes of fever & neutropenia
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2015-10; Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Clinically documented infection e.g., pneumonia, gastroenteritis, meningitis, septicemia, etc. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Recovery from fever neutropenia episode OR occurrence of clinically documented infection

SECONDARY OUTCOMES:
Death as a complication for infections | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Recovery from fever & neutropenia OR death as a complication of severe infection

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Kern WV. Risk assessment and risk-based therapeutic strategies in febrile neutropenia. Curr Opin Infect Dis. 2001 Aug;14(4):415-22. doi: 10.1097/00001432-200108000-00003. PMID 11964858
- [Background] Klastersky J, Paesmans M, Georgala A, Muanza F, Plehiers B, Dubreucq L, Lalami Y, Aoun M, Barette M. Outpatient oral antibiotics for febrile neutropenic cancer patients using a score predictive for complications. J Clin Oncol. 2006 Sep 1;24(25):4129-34. doi: 10.1200/JCO.2005.03.9909. PMID 16943529
- [Background] Klastersky J, Paesmans M, Rubenstein EB, Boyer M, Elting L, Feld R, Gallagher J, Herrstedt J, Rapoport B, Rolston K, Talcott J. The Multinational Association for Supportive Care in Cancer risk index: A multinational scoring system for identifying low-risk febrile neutropenic cancer patients. J Clin Oncol. 2000 Aug;18(16):3038-51. doi: 10.1200/JCO.2000.18.16.3038. PMID 10944139
- [Background] Kleinberg M, Bow EJ. Introduction: Approach to the Patient. In Kleinberg M (ed) Managing Infections in Patients With Hematological Malignancies. Humana Press 2010; 1-12
- [Background] Rolston KV. Risk assessment and risk-based therapy in febrile neutropenic patients. Eur J Clin Microbiol Infect Dis. 1998 Jul;17(7):461-3. doi: 10.1007/BF01691127. No abstract available. PMID 9764547
- [Background] Rolston KI, Bodey G. Management of the Neutropenic Patient with Fever. In Safdar A (ed) Principles and Practice of Cancer Infectious Diseases. Humana Press 2011; 95-103.
- [Background] Talcott JA, Finberg R, Mayer RJ, Goldman L. The medical course of cancer patients with fever and neutropenia. Clinical identification of a low-risk subgroup at presentation. Arch Intern Med. 1988 Dec;148(12):2561-8. PMID 3196123
- [Background] Talcott JA, Siegel RD, Finberg R, Goldman L. Risk assessment in cancer patients with fever and neutropenia: a prospective, two-center validation of a prediction rule. J Clin Oncol. 1992 Feb;10(2):316-22. doi: 10.1200/JCO.1992.10.2.316. PMID 1732432